CLINICAL TRIAL: NCT02085720
Title: Prevalence of Obstructive Sleep Apnea Syndrome and CPAP Adherence in the Elderly Chinese Population
Brief Title: Prevalence of OSAS in Chinese Elderly and Its CPAP Compliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Susanna SS Ng, Specialist, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Elderly OSA/Ng/2011
Record Dates: First submitted 2014-03-07; First posted 2014-03-13 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-03

CONDITIONS: Obstructive Sleep Apnea Syndrome; Restless Leg Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Restless Legs Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chinese elderly OSAS (Experimental): Subjects will be recruited in the community elderly center with home sleep study done. Those with significant OSAS will be prescribed with CPAP therapy and subsequent compliance is monitored.
  Interventions: Device: CPAP therapy

INTERVENTIONS:
Device: CPAP therapy — As OSA may increase the risk of cardiovascular mortality, all elderly subjects with AHI ≥ 15 or those with AHI ≥ 5 plus either cardiovascular risk factors or ESS score ≥ 10 received patient education program. Elderly subjects who agree for home CPAP treatment were prescribed nasal CPAP units with time clocks to assess objective compliance (run time). ESS, sleep apnea specific quality of life index (SAQLI), and cognitive function tests were performed at baseline, 3 months, 6 months and 12 months after CPAP treatment.

SUMMARY:
Objective: Obstructive sleep apnoea syndrome (OSAS) is a common form of sleep-disordered breathing (SDB) causing sleep fragmentation, daytime sleepiness, cognitive function impairment, and poor health status in addition to increased risk of cardiovascular complications. OSAS is equally common among the middle-aged male Caucasian and Hong Kong (HK) Chinese populations with a prevalence of at least 4%. However, the prevalence of OSAS in the elderly population in Asia including HK is unknown.

Study Design: A sleep questionnaire will be conducted for 1000 subjects aged at least 60 yrs in the elderly community centers focusing on symptoms of OSAS, subjective sleepiness, restless leg syndrome, and sleep-related habits and routines, in addition to past medical history and medications. Home sleep study (EMBLETTA) capable of recording sleep (a single EEG channel), respiratory events, snoring, respiratory efforts and oximetry will be performed on 300 subjects randomly. Those who have negative or technical inadequate EMBLETTA study with a high pre-test probability of moderate to severe OSA will be invited to undergo hospital-based polysomnography for confirmation of their sleep apnoea status. Subjects with AHI>15/hr regardless of symptoms or those with AHI 5-15/hr plus comorbid conditions or excessive daytime sleepiness will be offered continuous positive airway pressure (CPAP) titration followed by CPAP treatment, with serial assessment of subjective sleepiness, quality of life, and cognitive function.

Outcome measures: the prevalence rates of SDB (AHI>10, >15 and >30/hr), OSAS, and other sleep disturbances, such as restless leg syndrome (RLS). In addition, we will examine the factors which are predictive of the presence of SDB in this population, and assess the CPAP acceptance, compliance, and treatment outcome of those with OSAS.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is a common form of sleep-disordered breathing (SDB) characterized by repetitive episodes of cessation of breathing during sleep due to upper airway collapse. It causes sleep fragmentation, disabling daytime sleepiness, impaired cognitive function and poor quality of life. In addition, OSAS is associated with non-fatal and fatal cardiovascular consequences including sudden death, in addition to an increased risk of road traffic accidents. OSAS is equally common among the middle-aged male Caucasian and Hong Kong (HK) Chinese populations with a prevalence of at least 4%. However, the prevalence of OSAS in the elderly in Southeast Asia is unknown. Sleep disturbances, such as daytime sleepiness, SDB and non-respiratory causes including insomnia, restless leg syndrome are common in the elderly. There are also more frequent and sometimes prolonged nocturnal awakenings, leading to a decline in sleep efficiency (total time asleep as percentage of time in bed). However, the disruption of sleep architecture can be exaggerated by the presence of OSAS. The associated hypersomnolence can exacerbate the normal tendency in older people to sleep during the day, affecting their functional independence.

While OSAS produces large negative impacts on health and quality of life, the recognition is not always straightforward because of the presence of co-morbidities and normal age-related changes in sleep quality and behavior. Once OSAS is suspected, it is not only relatively easy to diagnose, but usually responds well to treatment with CPAP.

Method A sleep questionnaire will be conducted for 1000 subjects aged at least 60 yrs in the elderly community centers focusing on symptoms of OSAS, subjective sleepiness, restless leg syndrome, and sleep-related habits and routines, in addition to past medical history and medications. Home sleep study with the EMBLETTA device capable of recording sleep (a single EEG channel), respiratory events, snoring, respiratory efforts and oximetry will be performed on 300 subjects randomly. Descriptions of the device and the validity of the methods used to collect and display data have been published previously among both local Chinese and other populations. It is a multi-channel screening tool that measures airflow through a nasal cannula connected to a pressure transducer, providing an AHI based on recording time. It also detects both respiratory and abdominal efforts through the effort sensor and can differentiate between obstructive and central events. The body position is detected by the built-in sensors. Respiratory events are scored when desaturations of at least 4% occurred in the absence of moving artifacts and irrespective of co-existing changes in snoring or heart rate. A hypopnea is defined as a decrease in airflow by 50% of baseline for at least 10 seconds. Data are included in the analysis if the total recorded evaluation time of 4 hrs or longer is obtained during the EMBLETTA study.

Those who have negative or technical inadequate EMBLETTA study with a high pre-test probability of moderate to severe OSA will be invited to undergo hospital-based polysomnography for confirmation of their sleep apnoea status.

As OSA may increase the risk of cardiovascular mortality, all elderly subjects with AHI ≥ 15 or those with AHI ≥ 5 plus either cardiovascular risk factors or Epworth Sleepiness Score (ESS) score ≥ 10 received patient education program. Subjects who agreed for CPAP therapy were offered basic CPAP education package consisting of a 10-min CPAP education programme by a respiratory nurse explaining the basic operation and care of the CPAP device and the mask, educational brochure on OSA and CPAP treatment in Chinese, and careful mask fitting, and a short trial of CPAP therapy with the an automatic CPAP machine (AUTOSET CPAP) device (RESMED, Sydney, Australia) for approximately 30 minutes for acclimatization in the afternoon. Attended CPAP titration will be performed with the AUTOSET auto-titrating device in our hospital. Throughout the night and the next morning the nurses on duty would deal with any discomfort related to the CPAP treatment. The CPAP pressure for each patient will be set at the minimal pressure needed to abolish snoring, obstructive respiratory events and airflow limitation for 95% of the night as determined by the overnight AutoSet CPAP titration study. The patients subsequently will be followed up by physicians and nurses at the CPAP clinic in 1 month and 3 months later to deal with any problem with the CPAP device or mask fit. Subjects who agreed for home CPAP treatment will be prescribed nasal CPAP units with time clocks to assess objective compliance (run time). ESS, sleep apnea-specific quality of life index (SAQLI), and cognitive function tests will be performed at baseline and at 3 months after CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 60 years
* able to give consent

Exclusion Criteria:

* none

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 819 (Actual)
Dates: Start 2007-09; Primary Completion 2010-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanna SS Ng, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Community centers for elderly, Hong Kong, Hong Kong SAR, Hong Kong

REFERENCES:
- [Background] Engleman HM, Douglas NJ. Sleep. 4: Sleepiness, cognitive function, and quality of life in obstructive sleep apnoea/hypopnoea syndrome. Thorax. 2004 Jul;59(7):618-22. doi: 10.1136/thx.2003.015867. PMID 15223874
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Barcelo A, Pierola J, de la Pena M, Esquinas C, Sanchez-de la Torre M, Ayllon O, Alonso A, Agusti AG, Barbe F. Day-night variations in endothelial dysfunction markers and haemostatic factors in sleep apnoea. Eur Respir J. 2012 Apr;39(4):913-8. doi: 10.1183/09031936.00039911. Epub 2011 Aug 18. PMID 21852330
- [Background] Masa JF, Rubio M, Findley LJ. Habitually sleepy drivers have a high frequency of automobile crashes associated with respiratory disorders during sleep. Am J Respir Crit Care Med. 2000 Oct;162(4 Pt 1):1407-12. doi: 10.1164/ajrccm.162.4.9907019. PMID 11029353
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Bearpark H, Elliott L, Grunstein R, Cullen S, Schneider H, Althaus W, Sullivan C. Snoring and sleep apnea. A population study in Australian men. Am J Respir Crit Care Med. 1995 May;151(5):1459-65. doi: 10.1164/ajrccm.151.5.7735600.
- [Background] Ip MS, Lam B, Lauder IJ, Tsang KW, Chung KF, Mok YW, Lam WK. A community study of sleep-disordered breathing in middle-aged Chinese men in Hong Kong. Chest. 2001 Jan;119(1):62-9. doi: 10.1378/chest.119.1.62. PMID 11157585
- [Background] Feinsilver SH, Hertz G. Sleep in the elderly patient. Clin Chest Med. 1993 Sep;14(3):405-11. PMID 8222559
- [Background] Hume KI, Van F, Watson A. A field study of age and gender differences in habitual adult sleep. J Sleep Res. 1998 Jun;7(2):85-94. doi: 10.1046/j.1365-2869.1998.00103.x. PMID 9682179
- [Background] Ng SS, Chan TO, To KW, Ngai J, Tung A, Ko FW, Hui DS. Validation of Embletta portable diagnostic system for identifying patients with suspected obstructive sleep apnoea syndrome (OSAS). Respirology. 2010 Feb;15(2):336-42. doi: 10.1111/j.1440-1843.2009.01697.x. PMID 20199644
- [Background] Dingli K, Coleman EL, Vennelle M, Finch SP, Wraith PK, Mackay TW, Douglas NJ. Evaluation of a portable device for diagnosing the sleep apnoea/hypopnoea syndrome. Eur Respir J. 2003 Feb;21(2):253-9. doi: 10.1183/09031936.03.00298103. PMID 12608438
- [Background] Hui DS, Chan JK, Choy DK, Ko FW, Li TS, Leung RC, Lai CK. Effects of augmented continuous positive airway pressure education and support on compliance and outcome in a Chinese population. Chest. 2000 May;117(5):1410-6. doi: 10.1378/chest.117.5.1410. PMID 10807830
- [Background] Flemons WW, Reimer MA. Development of a disease-specific health-related quality of life questionnaire for sleep apnea. Am J Respir Crit Care Med. 1998 Aug;158(2):494-503. doi: 10.1164/ajrccm.158.2.9712036. PMID 9700127

RESULTS

PARTICIPANT FLOW:
Groups:
- Chinese Elderly OSAS: We conducted a sleep questionnaire survey among the elders aged 60 years or more in the community centres followed by level 3 home sleep study (EMBLETTA). Subjects with an apnea hypopnea index (AHI) ≥ 15 alone and those with AHI ≥ 5 plus either cardiovascular risk factors or Epworth Sleepiness Score (ESS) ≥ 10 were offered continuous positive airway pressure (CPAP) treatment.
  CPAP therapy: Elderly subjects who agreed for home CPAP treatment were prescribed nasal CPAP units with time clocks to assess objective compliance (run time). Epworth Sleepiness Score (ESS), sleep apnea specific quality of life index (SAQLI), and cognitive function tests were performed at baseline, 3 months, 6 months and 12 months after CPAP treatment.
Period: Overall Study
Arm/Group | Chinese Elderly OSAS
Started | 819
Completed | 819
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chinese Elderly OSAS
Number analyzed (Participants) | 819
Age, Continuous [Mean (Standard Deviation); unit: years]
  Total | 73.9 (7.5)
  Men | 73.4 (6.9)
  Female | 74.1 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 612
  Male | 207
Region of Enrollment [Number; unit: participants]
  Hong Kong | 819
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2]
  Total | 24.2 (3.6)
  Men | 24.3 (3.3)
  Female | 24.2 (3.7)
Neck circumference [Mean (Standard Deviation); unit: cm]
  Total | 34.9 (3.4)
  Men | 37.7 (2.9)
  Female | 33.8 (2.9)
Smoking status [Number; unit: participants]
  Non smoker | 696
  Smoker | 123
Alcohol drinker [Number; unit: participants]
  Non drinker | 630
  drinker | 189
Epworth Sleepiness Score [Mean (Standard Deviation); unit: units on a scale] — The ESS questionnaire is specific to symptoms of daytime sleepiness and subjects are asked to score the likelihood of falling asleep in eight different situations with different levels of stimulation, adding up to a total score of 0-24. The higher the score, the sleepy the subject is in the daytime. Usually the cut off of 10 is used to indicate abnormal sleepiness than usual.
  units on a scale
    Total | 6.6 (5.2)
    Men | 7.0 (5.2)
    Female | 6.5 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Obstructive Sleep Apnea Syndrome in Chinese Elderly
Description: Subjects who have completed the questionnaires and consented for sleep study are invited to undergo a portable at-home sleep study (EMBLETTA). It is a multi-channel screening tool that measures airflow through a nasal cannula connected to a pressure transducer, providing an apnea hypopnea index (AHI) based on recording time. AHI is the average number of events per hour while 5-15 events per hour denotes mild OSA, 16-30 events moderate OSA, and >30 events severe OSA. Obstructive sleep apnea syndrome is defined as AHI 15 events or above or AHI being 5 or above pulus ESS 10 or more. This measure is reporting the percentage of participants with OSAS.
Time Frame: 3 years
Measure: Number; unit: % of participants
Arm/Group | Chinese Elderly OSAS
Number analyzed (Participants) | 819
% of participants | 15
Statistical Analysis 1: Comparison: Chinese Elderly OSAS; Test type: Non-Inferiority or Equivalence — Data were given as means and standard deviations, unless otherwise stated. AHI was categorized as ≥ 5, ≥ 10, ≥ 15 and ≥ 20. The frequency distribution of responses on the SHQ and their relationship to AHI was assessed with the chi-squared analysis. The association of variables such as age, BMI, neck circumference, ESS and sleep health questionnaire responses versus AHI was evaluated using one-way analysis of variance and Pearson Correlation Analysis; p < 0.05, ANOVA

2. Secondary Outcome: Prevalence of Restless Leg Syndrome (RLS)
Description: RLS is a disorder characterized by disagreeable leg sensations that usually occur before sleep onset, causing an almost irresistible urge to move the legs. As minimal criteria for diagnosis, the following four features were required: (1) desire to move the extremities, often associated with paresthesias and/or dysesthesias; (2) motor restlessness; (3) worsening of symptoms at rest, with at least temporary relief by activity; and (4) worsening of symptoms in the evening or at night.
Time Frame: 3 years
Measure: Number; unit: % of participants
Groups:
- Chinese Elderly OSAS: RLS is a disorder characterized by disagreeable leg sensations that usually occur before sleep onset, causing an almost irresistible urge to move the legs. As minimal criteria for diagnosis, the following four features were required: (1) desire to move the extremities, often associated with paresthesias and/or dysesthesias; (2) motor restlessness; (3) worsening of symptoms at rest, with at least temporary relief by activity; and (4) worsening of symptoms in the evening or at night.
Arm/Group | Chinese Elderly OSAS
Number analyzed (Participants) | 819
% of participants | 13.8

3. Secondary Outcome: CPAP Compliance Among Chinese Elderly
Description: Elderly subjects who agree for home CPAP treatment are prescribed nasal CPAP units with time clocks to assess objective compliance (run time).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Chinese Elderly OSAS
Number analyzed (Participants) | 30
hours | 4.2 (2.2)

4. Secondary Outcome: AHI Result
Time Frame: 1 year
Measure: Number; unit: % of participants
Groups:
- AHI Result: Subjects who had completed the questionnaires and consented for sleep study were invited to undergo a portable at-home sleep study. In the afternoon, subjects attended the pulmonary function laboratory to be fitted with the EmblettaTM portable diagnostic system (PDS, Medcare, Iceland). It is a multi-channel screening tool that measures airflow through a nasal cannula connected to a pressure transducer, providing an AHI based on recording time. It also detects both respiratory and abdominal efforts through the effort sensor and can differentiate between obstructive and central events. Respiratory events were scored when desaturations of at least 4% occurred in the absence of moving artifacts and irrespective of co-existing changes in snoring or heart rate. A hypopnea was defined as a decrease in airflow by 50% of baseline for at least 10 seconds. Data were included in the analysis if the total recorded evaluation time of 4 hrs or longer was obtained during the EmblettaTM PDS study.
Arm/Group | AHI Result
Number analyzed (Participants) | 234
% of participants
  AHI >/5 | 66.7
  AHI >/10 | 43.6
  AHI >/15 | 29.9
  AHI >/20 | 19.2

5. Secondary Outcome: Sleep and Health Questionnaire Result
Time Frame: 1 year
Measure: Number; unit: % of participants
Groups:
- Sleep Heatlh Questionnaire Result: We conducted a sleep questionnaire survey among the elders aged 60 years or more in the community centres.
Arm/Group | Sleep Heatlh Questionnaire Result
Number analyzed (Participants) | 819
% of participants
  Impaired performance ability (mild) | 41.5
  Impaired performance ability (moderate) | 8.5
  Impaired performance ability | 8.7
  Sleepiness interfered with daily tasks (mild) | 10.2
  Sleepiness interfered with daily tasks (moderate) | 3.4
  Sleepiness interfered with daily tasks(severe) | 3.8
  Impaired energy level (mild) | 39.2
  Impaired energy level (moderate) | 8.0
  Impaired energy level (severe) | 9.4
  Daytime sleepiness (mild) | 41.1
  Daytime sleepiness (moderate) | 8.5
  Daytime sleepiness (severe) | 22.8
  Snoring intensity (past month) (mild) | 33.0
  Snoring intensity (past month) (moderate) | 8.2
  Snoring intensity (past month) (severe) | 5.1
  Frequent awakenings (mild) | 38.3
  Frequent awakenings (moderate) | 8.6
  Frequent awakenings (severe) | 19.3
  Difficulty falling asleep (mild) | 48.4
  Difficulty falling asleep (moderate) | 7.8
  Difficulty falling asleep (severe) | 9.9
  observed awakenings (mild) | 6.6
  observed awakenings (moderate) | 0.7
  observed awakenings (severe) | 0.8
  observed choking (mild) | 2.8
  observed choking (moderate) | 1.1
  observed choking (severe) | 0.7
  Observed apnea (mild) | 1.7
  Observed apnea (moderate) | 0.4
  Observed apnea (severe) | 0.6

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Chinese Elderly OSAS
Serious Adverse Events (participants affected / at risk) | 0/819
Other Adverse Events (participants affected / at risk) | 0/819

LIMITATIONS AND CAVEATS:
Subjects were chosen from the community centers and it is possible that those with more symptoms would be more eager to join the study; mre females than males; those who participated in the home sleep study were younger, with slightly higher ESS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No